CLINICAL TRIAL: NCT01345929
Title: A Multicenter, Double-Blind, Randomized, Phase 3 Study to Compare the Safety and Efficacy of Intravenous CXA-201 and Intravenous Levofloxacin in Complicated Urinary Tract Infection, Including Pyelonephritis
Brief Title: Study Comparing the Safety and Efficacy of Intravenous CXA-201 and Intravenous Levofloxacin in Complicated Urinary Tract Infection, Including Pyelonephritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7625A-005; CXA-cUTI-10-04 (Other: Cubist Study Number); CXA-cUTI-10-05 (Other: Cubist Study # for Study 7625A-006); NCT01345955 (obsolete NCT alias)
Record Dates: First submitted 2011-04-28; First posted 2011-05-02 (Estimated); Results first posted 2015-01-15 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-09

CONDITIONS: Complicated Urinary Tract Infection; Pyelonephritis
Keywords: cUTI
MeSH Terms: conditions — Pyelonephritis | interventions — Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CXA-201 as treatment for cUTI (Experimental): CXA-201 IV infusion (1500mg q8) for 7 days
  Interventions: Drug: CXA-201
- Levofloxacin as treatment for cUTI (Active Comparator): Levofloxacin IV infusion (750mg qd) for 7 days
  Interventions: Drug: Levofloxacin

INTERVENTIONS:
Drug: CXA-201 — CXA-201 IV infusion (1500mg q8) for 7 days
  Arms: CXA-201 as treatment for cUTI
Drug: Levofloxacin — Levofloxacin IV infusion (750mg qd) for 7 days
  Arms: Levofloxacin as treatment for cUTI

SUMMARY:
This is a Phase 3, multicenter, prospective, randomized, double-blind, double dummy study of CXA 201 IV infusions (1500 mg q8h) versus levofloxacin IV infusions (750 mg qd) for the treatment of adults with a cUTI (including pyelonephritis).

DETAILED DESCRIPTION:
Approximately 500 subjects will be enrolled into this study and randomized 1:1 to receive CXA-201 or comparator (levofloxacin) resulting in 250 subjects per treatment arm. Subject participation will require a minimum commitment of 35 days and a maximum of 42 days. Subjects will be hospitalized for the administration of all doses of IV study therapy. A test of cure visit will occur at 7 days after the last dose of study drug and a late follow-up evaluation or contact will occur a minimum of 28 days and a maximum of 35 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to any study-related procedure not part of normal medical care (a legally acceptable representative may provide consent if the subject is unable to do so, provided this is approved by local country and institution specific guidelines).
2. Be males or females ≥ 18 years of age
3. If female, subject is non-lactating, and is either:

   1. Not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile due to bilateral tubal ligation, bilateral oophorectomy, or hysterectomy; or
   2. Of childbearing potential and is practicing a barrier method of birth control (e.g., a diaphragm or contraceptive sponge) along with 1 of the following methods: oral or parenteral contraceptives (for 3 months prior to study drug administration), or a vasectomized partner. Or, subject is practicing abstinence from sexual intercourse. Subjects must be willing to practice these methods for the duration of the trial and for at least 35 days after last dose of study medication.
4. Males are required to practice reliable birth control methods (condom or other barrier device) during the conduct of the study and for at least 35 days after last dose of study medication.
5. Pyuria (white blood cell [WBC] count > 10/μL in unspun urine or ≥ 10 per high power field in spun urine).
6. Clinical signs and/or symptoms of cUTI, either of:

   1. Pyelonephritis, as indicated by at least 2 of the following:

      * Documented fever (oral temperature > 38°C) accompanied by patient symptoms of rigors, chills, or "warmth";
      * Flank pain;
      * Costovertebral angle tenderness or suprapubic tenderness on physical exam; or
      * nausea or vomiting; OR
   2. Complicated lower UTI, as indicated by at least 2 of the following:

      * At least 2 of the following new or worsening symptoms of cUTI:

        * Dysuria; urinary frequency or urinary urgency;
        * Documented fever (oral temperature > 38°C) accompanied by patient symptoms of rigors, chills, or "warmth";
        * Suprapubic pain or flank pain;
        * Costovertebral angle tenderness or suprapubic tenderness on physical exam; or
        * Nausea or vomiting; plus,
      * At least 1 of the following complicating factors:

        * Males with documented history of urinary retention;
        * Indwelling urinary catheter that is scheduled to be removed during IV study therapy and before the EOT;
        * Current obstructive uropathy that is scheduled to be medically or surgically relieved during IV study therapy and before the EOT; or
        * Any functional or anatomical abnormality of the urogenital tract (including anatomic malformations or neurogenic bladder) with voiding disturbance resulting in at least 100 mL residual urine.
7. Have a pretreatment baseline urine culture specimen obtained within 24 hours before the start of administration of the first dose of study drug.

   NOTE: Subjects may be enrolled in this study and start IV study drug therapy before the Investigator knows the results of the baseline urine culture.
8. Require IV antibacterial therapy for the treatment of the presumed cUTI.

Exclusion Criteria:

1. Have a documented history of any moderate or severe hypersensitivity or allergic reaction to any β-lactam or quinilone antibacterial (Note: for β-lactams, a history of a mild rash followed by uneventful re-exposure is not a contraindication to enrollment)
2. Have a concomitant infection at the time of randomization, which requires non-study systemic antibacterial therapy in addition to IV study drug therapy. (Drugs with only gram-positive activity [e.g., vancomycin, linezolid] are allowed.)
3. Receipt of any amount of potentially therapeutic antibacterial therapy after collection of the pretreatment baseline urine culture and before administration of the first dose of study drug.
4. Receipt of any dose of a potentially therapeutic antibacterial agent for the treatment of the current UTI within 48 hours before the study-qualifying pretreatment baseline urine is obtained (exceptions: subjects with an active cUTI who have received prior antibiotics may be enrolled provided a minimum of 48 hours have elapsed between the last dose of the prior antibiotic and the time of obtaining the baseline urine specimen. Subjects receiving current antibiotic prophylaxis for cUTI who present with signs and symptoms consistent with an active new cUTI may be enrolled provided all other eligibility criteria are met including obtaining a pre-treatment qualifying baseline urine culture).
5. Intractable urinary infection at baseline that the Investigator anticipates would require more than 7 days of study drug therapy.
6. Complete, permanent obstruction of the urinary tract.
7. Confirmed fungal urinary tract infection at time of randomization (with ≥ 103 fungal CFU/mL).
8. Permanent indwelling bladder catheter or urinary stent including nephrostomy.
9. Suspected or confirmed perinephric or intrarenal abscess.
10. Suspected or confirmed prostatitis.
11. Ileal loop or known vesico-ureteral reflux.
12. Severe impairment of renal function including an estimated CrCl < 30 mL/min, requirement for peritoneal dialysis, hemodialysis or hemofiltration, or oliguria (< 20 mL/h urine output over 24 hours).
13. Current urinary catheter that is not scheduled to be removed before the EOT (intermittent straight catheterization during the IV study drug administration period is acceptable).
14. Any condition or circumstance that, in the opinion of the Investigator, would compromise the safety of the subject or the quality of study data.
15. Any rapidly progressing disease or immediately life-threatening illness including acute hepatic failure, respiratory failure, and septic shock.
16. Immunocompromising condition, including established AIDS, hematological malignancy, or bone marrow transplantation, or immunosuppressive therapy including cancer chemotherapy, medications for prevention of organ transplantation rejection, or the administration of corticosteroids equivalent to or greater than 40 mg of prednisone per day administered continuously for more than 14 days preceding randomization.
17. One or more of the following laboratory abnormalities in baseline specimens: aspartate aminotransferase (AST [SGOT]), alanine aminotransferase (ALT [SGPT]), alkaline phosphatase, or total bilirubin level greater than 3 times the upper limit of normal (ULN), absolute neutrophil count less than 500/μL, platelet count less than 40,000/μL, or hematocrit less than 20%.
18. Participation in any clinical study of an investigational product within 30 days prior to the proposed first day of study drug.
19. Previous participation in any study of CXA-101 or CXA-201.
20. Women who are pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2011-06-20 (Actual); Primary Completion 2013-08-11 (Actual); Study Completion 2013-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Obiamiwe Umeh, M.D., MSc., Study Director — Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (76):
- United States (5):
  - San Diego, California
  - Wheat Ridge, Colorado
  - Hialeah, Florida
  - Teaneck, New Jersey
  - Charleston, South Carolina
- Brazil (7):
  - Belo Horizonte, Minas Gerais
  - Porto Alegre, Rio Grande de Sul
  - Joinville, Santa Catarina
  - Campinas, São Paulo
  - Sao Jose de Rio Preto, São Paulo
  - Rio de Janeiro
  - São Paulo
- Colombia (4):
  - Cali, Valle del Cauca Department
  - Armenia
  - Barranquilla
  - Bogotá
- Estonia (3):
  - Kohtla-Järve
  - Tallinn
  - Tartu
- Tbilisi, Georgia
- Germany (2):
  - Giessen, Hesse
  - Lübeck, Schleswig-Holstein
- Hungary (9):
  - Miskolc, Borsod-Abauj Zemplen county
  - Gyor, Budapest
  - Szentes, Csongrád megye
  - Sopron, Győr-Moson-Sopron
  - Salgótarján, Nógrád megye
  - Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Zalaegerszeg, Zala County
  - Budapest
  - Tatabánya
- Israel (6):
  - Kfar Saba, Sharon
  - Petah Tikva, Teah Tiqwa
  - Tel Litwinsky, Tel Aviv
  - Haifa
  - Jerusalem
  - Safed
- Latvia (5):
  - Daugavpils
  - Liepāja
  - Riga
  - Valmiera
  - Ventspills
- Mexico (4):
  - Guadalajara, Jalisco
  - Chihuahua City
  - San Luis Potosí City
  - Veracruz
- Chisinau, Moldova
- Romania (7):
  - Oradea, Bihor County
  - Bucharest, București
  - Timișoara, Timiș County
  - Brasov
  - Bucharest
  - Iași
  - Sibiu
- Russia (7):
  - Kemerovo
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Penza
  - Saint Petersburg
  - Saratov
- Belgrade, Serbia
- Slovakia (5):
  - Banská Bystrica
  - Levice
  - Martin
  - Prešov
  - Skalica
- South Africa (5):
  - Bloemfontein, Free State
  - Pretoria, Gauteng
  - Soweto, Gauteng
  - Middleburg, Mpumalanga
  - Bellville, Western Cape
- Thailand (4):
  - Nakorn Ratchasima, Changwat Nakhon Ratchasima
  - Chiang Mai
  - Lopburi
  - Prachuap Khiri Khan

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Popejoy MW, Long J, Huntington JA. Analysis of patients with diabetes and complicated intra-abdominal infection or complicated urinary tract infection in phase 3 trials of ceftolozane/tazobactam. BMC Infect Dis. 2017 May 2;17(1):316. doi: 10.1186/s12879-017-2414-9. PMID 28464828
- [Derived] Xiao Y, Tong ML, Liu LL, Lin LR, Chen MJ, Zhang HL, Zheng WH, Li SL, Lin HL, Lin ZF, Xing HQ, Niu JJ, Yang TC. Novel predictors of neurosyphilis among HIV-negative syphilis patients with neurological symptoms: an observational study. BMC Infect Dis. 2017 Apr 26;17(1):310. doi: 10.1186/s12879-017-2339-3. PMID 28446129
- [Derived] Kullar R, Wagenlehner FM, Popejoy MW, Long J, Yu B, Goldstein EJ. Does moderate renal impairment affect clinical outcomes in complicated intra-abdominal and complicated urinary tract infections? Analysis of two randomized controlled trials with ceftolozane/tazobactam. J Antimicrob Chemother. 2017 Mar 1;72(3):900-905. doi: 10.1093/jac/dkw486. PMID 27999024
- [Derived] Armstrong ES, Mikulca JA, Cloutier DJ, Bliss CA, Steenbergen JN. Outcomes of high-dose levofloxacin therapy remain bound to the levofloxacin minimum inhibitory concentration in complicated urinary tract infections. BMC Infect Dis. 2016 Nov 25;16(1):710. doi: 10.1186/s12879-016-2057-2. PMID 27887579
- [Derived] Huntington JA, Sakoulas G, Umeh O, Cloutier DJ, Steenbergen JN, Bliss C, Goldstein EJ. Efficacy of ceftolozane/tazobactam versus levofloxacin in the treatment of complicated urinary tract infections (cUTIs) caused by levofloxacin-resistant pathogens: results from the ASPECT-cUTI trial. J Antimicrob Chemother. 2016 Jul;71(7):2014-21. doi: 10.1093/jac/dkw053. Epub 2016 Mar 18. PMID 26994090
- [Derived] Wagenlehner FM, Umeh O, Steenbergen J, Yuan G, Darouiche RO. Ceftolozane-tazobactam compared with levofloxacin in the treatment of complicated urinary-tract infections, including pyelonephritis: a randomised, double-blind, phase 3 trial (ASPECT-cUTI). Lancet. 2015 May 16;385(9981):1949-56. doi: 10.1016/S0140-6736(14)62220-0. Epub 2015 Apr 27. PMID 25931244

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two P3 protocols were initiated (NCT01345929 and NCT01345955) subsequently, Cubist and FDA agreed that integrated data from the 2 protocols could be analyzed and reported in a single Clinical Study Report. A total of 1083 subjects were randomized to both arms, 558 to NCT01345929 and 525 to NCT01345955. Of these, 552 and 516 received treatment.
Groups:
- CXA-201 as Treatment for cUTI: CXA-201 IV infusion (1500mg q8) for 7 days
  CXA-201: CXA-201 IV infusion (1500mg q8) for 7 days
  Of the 1083 subjects in the integrated analysis set, 533 received CXA.
- Levofloxacin as Treatment for cUTI: Levofloxacin IV infusion (750mg qd) for 7 days
  Levofloxacin: Levofloxacin IV infusion (750mg qd) for 7 days
  Of the 1083 subjects in the integrated analysis set, 535 received levofloxacin.
Period: Overall Study
Arm/Group | CXA-201 as Treatment for cUTI | Levofloxacin as Treatment for cUTI
Started | 533 | 535
Completed | 512 | 516
Not Completed | 21 | 19
Not completed — Withdrawal by Subject | 9 | 8
Not completed — Lost to Follow-up | 9 | 9
Not completed — Adverse Event | 0 | 1
Not completed — Didn't meet eligibility criteria | 2 | 0
Not completed — 40,000 CFU/ML | 1 | 0
Not completed — Patient withdrawal | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CXA-201 as Treatment for cUTI | Levofloxacin as Treatment for cUTI | Total
Number analyzed (Participants) | 533 | 535 | 1068
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (19.52) | 48.6 (20.05) | 49.1 (19.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 374 | 380 | 754
  Male | 159 | 155 | 314

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Who Have Both a Per-subject Microbiological Outcome of Eradication and a Clinical Outcome of Cure at the Test of Cure (TOC) Visit in the Microbiological Modified ITT (mMITT) Population
Time Frame: Test of Cure Visit (7 Days [± 2 days] after completion of study drug administration)
Population: mMITT: Treated subjects, with baseline pathogen.
Measure: Number; unit: percentage of subjects
Arm/Group | CXA-201 as Treatment for cUTI | Levofloxacin as Treatment for cUTI
Number analyzed (Participants) | 398 | 402
percentage of subjects | 76.9 | 68.4
Statistical Analysis 1: Comparison: CXA-201 as Treatment for cUTI vs Levofloxacin as Treatment for cUTI; Test type: Non-Inferiority or Equivalence — Noninferiority was concluded if the lower bound of the 2-sided 95% CI was greater than -10%; Risk Difference (RD) = 8.5, 95% CI 2-sided [2.31 to 14.57]

2. Secondary Outcome: The Percentage of Subjects Who Have Both a Per-subject Microbiological Outcome of Eradication and a Clinical Outcome of Cure at the TOC Visit in the Microbiologically Evaluable (ME) Population.
Time Frame: Test of Cure Visit (7 Days [± 2 days] after completion of study drug administration)
Population: ME: Treated patients, with baseline pathogen, complied with protocol.
Measure: Number; unit: percentage of subjects
Arm/Group | CXA-201 as Treatment for cUTI | Levofloxacin as Treatment for cUTI
Number analyzed (Participants) | 341 | 353
percentage of subjects | 83.3 | 75.4
Statistical Analysis 1: Comparison: CXA-201 as Treatment for cUTI vs Levofloxacin as Treatment for cUTI; Test type: Non-Inferiority or Equivalence — Noninferiority was concluded if the lower bound of the 2-sided 95% CI was greater than -10%; Risk Difference (RD) = 8.0, 95% CI 2-sided [1.95 to 13.97]

ADVERSE EVENTS:
Arm/Group | CXA-201 as Treatment for cUTI | Levofloxacin as Treatment for cUTI
Serious Adverse Events (participants affected / at risk) | 15/533 | 18/535
Other Adverse Events (participants affected / at risk) | 108/533 | 101/535
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CXA-201 as Treatment for cUTI (N=533) | Levofloxacin as Treatment for cUTI (N=535)
Urinary tract infection (Infections and infestations) | 3 | 2
Pneumonia (Infections and infestations) | 2 | 0
Urosepsis (Infections and infestations) | 2 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 6
Emphysematous pyelonephritis (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Renal tubular acidosis (Renal and urinary disorders) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Diabetic retinopaty (Eye disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Hernia obstructive (General disorders) | 0 | 1
Contrast media allergy (Immune system disorders) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CXA-201 as Treatment for cUTI (N=533) | Levofloxacin as Treatment for cUTI (N=535)
Abdominal pain upper (Gastrointestinal disorders) | 7 | 6
Constipation (Gastrointestinal disorders) | 21 | 17
Diarrhoea (Gastrointestinal disorders) | 10 | 23
Nausea (Gastrointestinal disorders) | 15 | 9
Vomiting (Gastrointestinal disorders) | 6 | 6
Pyrexia (General disorders) | 8 | 4
Urinary tract infection (Infections and infestations) | 6 | 7
Alanine aminotransferase increased (Investigations) | 9 | 5
Aspartate aminotransferase increased (Investigations) | 9 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 4
Dizziness (Nervous system disorders) | 6 | 1
Headache (Nervous system disorders) | 31 | 26
Insomnia (Psychiatric disorders) | 7 | 14
Hypertension (Vascular disorders) | 16 | 7

LIMITATIONS AND CAVEATS:
Two identical P3 protocols were initiated (NCT01345929 and NCT01345955) subsequently, Cubist and FDA agreed that integrated data from the 2 protocols could be analyzed and reported in a single Clinical Study Report. These analyses are presented here.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator(s) must undertake not to submit any part of the data from this protocol for publication without the prior consent of Cubist Pharmaceuticals, Inc.